CLINICAL TRIAL: NCT02675829
Title: A Phase 2 Trial of Ado-Trastuzumab Emtansine for Patients With HER2 Amplified or Mutant Cancers
Brief Title: Trial of Ado-Trastuzumab Emtansine for Patients With HER2 Amplified or Mutant Cancers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-335
Record Dates: First submitted 2016-02-03; First posted 2016-02-05 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor Cancers; Lung Cancer; Bladder Cancer; Urinary Tract Cancers
Keywords: HER2 mutant; HER2 amplified; Ado-Trastuzumab Emtansine; 15-335
MeSH Terms: conditions — Lung Neoplasms; Urinary Bladder Neoplasms; Urologic Neoplasms | interventions — Ado-Trastuzumab Emtansine

ARMS (6):
- Cohort 1: Lung cancers, HER2 mutant (Experimental)
  Interventions: Drug: ado-trastuzumab emtansine
- Cohort 2: Lung cancers, HER2 amplified (Experimental)
  Interventions: Drug: ado-trastuzumab emtansine
- Cohort 3: Colorectal cancers (Experimental)
  Interventions: Drug: ado-trastuzumab emtansine
- Cohort 4: Endometrial cancers (Experimental)
  Interventions: Drug: ado-trastuzumab emtansine
- Cohort 5: Salivary gland cancers (Experimental)
  Interventions: Drug: ado-trastuzumab emtansine
- Cohort 6: Other solid cancers (Experimental)
  Interventions: Drug: ado-trastuzumab emtansine

INTERVENTIONS:
Drug: ado-trastuzumab emtansine — Ado-trastuzumab emtansine is administered intravenously at 3.6 mg/kg every 21 days (unless dose reduction and/or dose delays are required) until disease progression or unacceptable toxicity.

SUMMARY:
The purpose of this study is to find out what effects, a drug called ado-trastuzumab emtansine has on the patient and their cancer which is thought to be controlled by the abnormal HER2 gene.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are ≥18 years old.
* Pathologically confirmed advanced solid tumor cancers
* For Cohort 1, documented activating HER2 mutation in lung cancer by CLIA laboratory, specifically exon 20 insYVMA (Y772_A775dup), insGSP (G778_P780dup), insTGT (G776delinsVC), single base pair substitutions L755A, L755S, V777L, V659E, S310F, or another HER2 mutation approved by the Principal Investigator
* For Cohorts 2, 3, 4, 5, 6 documented HER2 amplification identified through next generation sequencing by MSK-IMPACT or at another Clinical Laboratory Improvement Amendments (CLIA) laboratory, or documented HER2 amplification by in-situ hybridization (ISH) with HER2/CEP17 ratio ≥2.0 at a CLIA laboratory. Patients with HER2 amplification identified by another method or criteria must be approved by the Principal Investigator and may enroll in the "Other" Cohort 4.
* Measurable or evaluable indicator lesion(s) as defined by RECIST v1.1. Patients without RECIST measurable disease will be eligible for enrollment to "Other" cohort provided their disease can be evaluated using another accepted response criteria (e.g. Gynecologic Cancer InterGroup (GCIG) CA125 Response Criteria, modified PET Response Criteria in Solid Tumors (PERCIST)). Patients with salivary gland cancers (Cohort 5) may be eligible on the basis of evaluable disease on modified PET.
* Karnofsky Performance Status 70% or above.
* Left ventricular ejection fraction (LVEF) ≥50% measured by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA).
* Negative β-human chorionic gonadotropin (hCG) pregnancy test within 2 weeks before enrollment for premenopausal women of reproductive capacity and for women less than 12 months after menopause. Pregnancy screening will be conducted for women up to the age of 50 years per institutional standard.
* Women of childbearing potential must agree to use of a highly effective method of contraception. Effective contraception is required during treatment and for 7 months following the last dose for female participants of reproductive potential and during treatment and for 4 months following the last dose for male participants with female sexual partners of reproductive potential. Male participants should also refrain from donating sperm during treatment and for 4 months following the last dose.
* Absolute neutrophil count ≥ 1,000/µL within 30 days prior to C1D1
* Platelet count ≥ 100,000/µL within 30 days prior to C1D1
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN), in case of Gilbert's syndrome, ≤ 2x ULN within 30 days prior to C1D1
* Aspartate aminotransferase and/or alanine aminotransferase ≤ 3 x ULN (≤ 5 x ULN if liver metastases are present) within 30 days prior to C1D1
* Provide written, informed consent to participate in the study and follow the study procedures

Exclusion Criteria:

* Prior therapy resulting in cumulative epirubicin dose ≥ 900mg/m2 or cumulative doxorubicin dose ≥ 500mg/m2 or equivalent dose of another anthracycline.
* Prior therapy with ado-trastuzumab emtansine (patients who had prior trastuzumab or other HER2 targeted agents are eligible).
* Symptomatic congestive heart failure (New York Heart Association Classification II-IV).
* Myocardial infarction or unstable angina within 6 months of enrollment.
* Unstable ventricular arrhythmia requiring treatment.
* Grade 3 or worse peripheral neuropathy as defined by CTCAE v4.1.
* Women who are pregnant or breast-feeding.
* Known hypersensitivity to any component of ado-trastuzumab emtansine.
* History of interstitial lung disease or pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
best overall response (ORR) | 2 years
  As soon as evaluations for each tumor assessment are completed, the Investigator should assess the patient's overall response (target plus non- target lesions) based on criteria and overall response algorithms as defined in RECIST version 1.1. Scans must be assessable for all evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Chaft, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

REFERENCES:
- [Derived] Mondaca S, Razavi P, Xu C, Offin M, Myers M, Scaltriti M, Hechtman JF, Bradley M, O'Reilly EM, Berger MF, Solit DB, Li BT, Abou-Alfa GK. Genomic Characterization of ERBB2-Driven Biliary Cancer and a Case of Response to Ado-Trastuzumab Emtansine. JCO Precis Oncol. 2019 Oct 17;3:PO.19.00223. doi: 10.1200/PO.19.00223. eCollection 2019. PMID 32923849
- [Derived] Li BT, Shen R, Buonocore D, Olah ZT, Ni A, Ginsberg MS, Ulaner GA, Offin M, Feldman D, Hembrough T, Cecchi F, Schwartz S, Pavlakis N, Clarke S, Won HH, Brzostowski EB, Riely GJ, Solit DB, Hyman DM, Drilon A, Rudin CM, Berger MF, Baselga J, Scaltriti M, Arcila ME, Kris MG. Ado-Trastuzumab Emtansine for Patients With HER2-Mutant Lung Cancers: Results From a Phase II Basket Trial. J Clin Oncol. 2018 Aug 20;36(24):2532-2537. doi: 10.1200/JCO.2018.77.9777. Epub 2018 Jul 10. PMID 29989854
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/